CLINICAL TRIAL: NCT00379327
Title: Acupuncture for Promotion of Timely Delivery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, John Farrar, MD, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AcuPTD-100
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2010-10

CONDITIONS: Delivery, Obstetric
Keywords: Pregnancy; Acupuncture; Pregnancy Outcome; Randomized Controlled Trial; Double-Blind Method
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real Accupuncture (Experimental): Acupuncture with a real needle that punctures the skin versus acupuncture needle that does not puncture the skin.
  Interventions: Procedure: Acupuncture
- Non-puncturing Acupuncture (Placebo Comparator): Acupuncture needle that touches but does not puncture the skin
  Interventions: Device: Non-puncturing Acupuncture Needle

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture administered in last three weeks of pregnancy
  Other Names: Asia Medicine Produces needle
  Arms: Real Accupuncture
Device: Non-puncturing Acupuncture Needle — Streitsberg non-Acupuncture Needle
  Other Names: Asia Medicine produces this needle
  Arms: Non-puncturing Acupuncture

SUMMARY:
The purpose of this study of 100 pregnant women is to determine if acupuncture using real needles that puncture the skin, starting at thirty seven weeks three days estimated gestational age (EGA), will increase the percentage of women delivering on or before the estimated date of confinement (EDC = 40 weeks EGA), compared with women treated identically but with placebo needles that do not puncture the skin.

DETAILED DESCRIPTION:
General Design This is a randomized controlled study of pregnant women to determine if acupuncture starting at thirty seven weeks three days EGA will increase the percentage of women delivering on or before the EDC, 40 weeks EGA.

The study participants will be recruited at three practices which utilize St. Francis Hospital in Wilmington Delaware, practices and hospital well known to the primary investigator. With the permission of the patients' physicians, charts of potentially eligible patients will be reviewed and eligible patients will be recruited into the study prior to 36 weeks EGA.

Upon enrollment, patients will be separated into nulliparous and parous groups and each group will be randomized into study intervention or control groups.

Of note, the candidate population is comprised of English and Spanish speakers. All invitational, explanatory, and consent materials and study instruments are available in both English and Spanish.

In addition to demographic information, initial and periodic "quality of life" and anxiety inventories will be administered. Based upon the current literature for applicability in this particular study population, the State-Trait Anxiety Index (STAI) and the Short Form 36 (SF-36) have been chosen as the test instruments.

Both primary care providers and enrolled patients will be asked every week to answer a single question with regards to whether or not they think the patient is receiving true or placebo acupuncture treatments. This will be done to analyze the efficacy of the blinding process.

At the time of enrollment, each patient will have a cervical exam performed by their physician to determine their individual baseline Bishop's Score. Subsequently, at each weekly obstetrical visit up to the patient's EDC, another cervical examination will be performed and a Bishop's Score obtained to assess cervical ripening.

Each subject will be seen twice weekly by the acupuncturist and will receive either actual acupuncture treatment or placebo (non-puncturing needles) treatment. Patients identified as "high risk" based upon the clinical judgment of the primary care physician will have external uterine pressure monitoring and fetal heart rate monitoring during the acupuncture treatments.

The acupuncture treatments will be administered in a standardized way by a single experienced medical acupuncturist certified by the state of Pennsylvania, to reduce the variability in the study. The acupuncture will be performed in a quiet area for all subjects. The newly validated and now commercially available placebo needle developed by Streitberger, et al will be used 34 and identical real needle using the same procedure for the placement of both types of needles. Briefly, a small bandage is applied to the skin covering a thin plastic disk over each acupuncture site. Either needle is placed through one of the small hole in the plastic portion of the bandage and through the underlying gauze. The sharp real needle easily penetrates the skin to the required depth, with no resistance imposed by the bandage. The blunt shaft of the placebo needle applies pressure on the skin as it retracts into the hollow handle, giving the appearance of the needle going into the skin. The bandage and gauze hold the placebo needle in place. The acupuncture needles will be manipulated for a few seconds on at the beginning and in the middle of the 30 minutes treatment period to try to elicit a sensation called the De qi. It is sometimes perceived by the subject as a dull ache that radiates from the point of insertion, or can be detected by the acupuncturist as a sense of increased resistance.

Since both the real and placebo needle groups reported feeling some sensation in Streitberger's validation study and the published study 35 blinding of the subject will be preserved. To ensure that the blinding is adequate, at each prenatal visit and at the postpartum follow up visit a simple question will be asked of study subjects and of their own physicians regarding which type of treatment (real versus placebo acupuncture) they believe the subject received in each session.

Primary Study Endpoints Our goal is to determine if our study intervention, acupuncture, will increase by 30% the number of women who have a timely delivery-- deliver on or before the EDC. Our study endpoint will be the EGA at the time of delivery. We will answer the question: "Was it a timely delivery?"

Primary Safety Endpoints If during the trial there is any evidence clinically or on monitor of uterine over-stimulation or fetal intolerance, the patient will remain enrolled as "intention to treat", but not continue with acupuncture treatments.

If the physician caring for the patient (obstetrician or FP-obstetrician) has any concerns that warrant the discontinuation of the acupuncture treatments, the patient will be withdrawn from the study and will be followed as "intention to treat".

ELIGIBILITY:
Inclusion Criteria:

1. A singleton pregnancy in cephalic presentation
2. Between 34 and 37 weeks gestation
3. Their pregnancy dating (due date) confirmed by at least one first or second trimester ultrasound
4. No fetal or maternal contraindications to vaginal delivery
5. No contraindication to carry to EDC (40w 0d)
6. Have the capacity to understand the requirements of the study

Exclusion Criteria:

1. Without adequate information of dating
2. High risk of Cesarean Delivery
3. Currently receiving acupuncture outside of study
4. Uncertainty of gestational age dating (according to the chart documentation)

Ages: 15 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2006-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
timely delivery -- deliver on or before the EDC

SECONDARY OUTCOMES:
State-Trait Anxiety Index, a self-administered questionnaire for assessment of anxiety
Short Form 36, a self-administered questionnaire for assessment of quality of life status
Modified Bishop's Score obtained to assess cervical ripening
Maternal and newborn outcomes

CONTACTS AND LOCATIONS:
Overall Officials: John T Farrar, MD, PhD, Study Director — University of Pennsylvania; Rebecca A Greenberg, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- St. Francis Hospital, Wilmington, Delaware, United States

REFERENCES:
- [Background] Caughey AB, Nicholson JM, Cheng YW, Lyell DJ, Washington AE. Induction of labor and cesarean delivery by gestational age. Am J Obstet Gynecol. 2006 Sep;195(3):700-5. doi: 10.1016/j.ajog.2006.07.003. PMID 16949399
- [Background] Caughey AB, Bishop JT. Maternal complications of pregnancy increase beyond 40 weeks of gestation in low-risk women. J Perinatol. 2006 Sep;26(9):540-5. doi: 10.1038/sj.jp.7211560. Epub 2006 Jul 13. PMID 16837930
- [Background] Rabl M, Ahner R, Bitschnau M, Zeisler H, Husslein P. Acupuncture for cervical ripening and induction of labor at term--a randomized controlled trial. Wien Klin Wochenschr. 2001 Dec 17;113(23-24):942-6. PMID 11802511
- [Background] Smith CA, Crowther CA. Acupuncture for induction of labour. Cochrane Database Syst Rev. 2004;(1):CD002962. doi: 10.1002/14651858.CD002962.pub2. PMID 14973999